CLINICAL TRIAL: NCT00405886
Title: A Randomised, Double-Blind, Placebo-Controlled, Clinical Dose-Ranging Trial to Evaluate Efficacy and Safety of a NMDA Antagonist for Oral Administration in Patients With Subjective Tinnitus
Brief Title: Neramexane for Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Dr. Matthias Zerm, Manager Public Disclosure, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ 92579-0508/1
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — neramexane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Neramexane 25mg/d (Experimental)
  Interventions: Drug: Neramexane
- Neramexane 50mg/d (Experimental)
  Interventions: Drug: Neramexane
- Neramexane 75mg/d (Experimental)
  Interventions: Drug: Neramexane
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neramexane — Oral tablets, duration: 16 weeks
  Arms: Neramexane 25mg/d; Neramexane 50mg/d; Neramexane 75mg/d
Drug: Placebo — Oral tablets, duration: 16 weeks
  Arms: Placebo

SUMMARY:
Tinnitus is commonly referred to as "ringing of the ears" - the perception of sounds in the absence of an external source of acoustic signals. Tinnitus may represent a severe disease and symptoms include depression, sleeping difficulties, decreased sound tolerance and hearing loss. One hypothesis is that tinnitus is caused by an increased activity of NMDA glutamate and dysfunctional alpha9/alpha10 acetylcholine receptors in the inner ear and central nervous system. Neramexane may alleviate tinnitus symptoms due to its NMDA and alpha9/alpha10 nACh receptor blocking activity. The purpose of this study is to assess the safety and efficacy of Neramexane compared with placebo in patients with subjective tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* main inclusion criterion: persistent, subjective, uni- or bilateral tinnitus

Exclusion Criteria:

* main exclusion criterion: intermittent or pulsatile tinnitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in tinnitus severity at the endpoint visit | Week 16
Comparison of adverse events (type, severity, seriousness, frequency, relatedness) between treatment arms | From baseline until week 20

CONTACTS AND LOCATIONS:
Overall Officials: Markus Suckfüll, MD PhD Ass. Prof., Study Chair — Ludwig-Maximilians - University of Munich
Locations (2):
- Vienna, Austria
- Munich, Germany

REFERENCES:
- [Result] Suckfull M, Althaus M, Ellers-Lenz B, Gebauer A, Gortelmeyer R, Jastreboff PJ, Moebius HJ, Rosenberg T, Russ H, Wirth Y, Krueger H. A randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of neramexane in patients with moderate to severe subjective tinnitus. BMC Ear Nose Throat Disord. 2011 Jan 11;11:1. doi: 10.1186/1472-6815-11-1. PMID 21223542
- [Derived] Gortelmeyer R, Schmidt J, Suckfull M, Jastreboff P, Gebauer A, Kruger H, Wittmann W. Assessment of tinnitus-related impairments and disabilities using the German THI-12: sensitivity and stability of the scale over time. Int J Audiol. 2011 Aug;50(8):523-9. doi: 10.3109/14992027.2011.578591. PMID 21751942